CLINICAL TRIAL: NCT07084740
Title: Study and Modeling of Perforator Flap Vascularization
Acronym: EMoVaLP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL25_0082; 2025-A00951-48 (Other: ANSM)
Record Dates: First submitted 2025-07-02; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Reconstructive Surgery Using Pedicled Perforating or Free Perforating Flaps; Pelvic Eschar; Traumatic Pathology of the Lower and/or Upper Limb
Keywords: Perforasome; perforator flap; PeriCam; Periflux EPOS; tissue perfusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PeriCam and PeriFlux measurements (Experimental): PeriCam and PeriFlux measurements
  Interventions: Diagnostic Test: PeriCam and PeriFlux measurements

INTERVENTIONS:
Diagnostic Test: PeriCam and PeriFlux measurements — PeriCam and PeriFlux measurements

SUMMARY:
The aim of reconstructive surgery is to restore physical integrity altered by trauma, congenital malformations or cancerous pathologies. Several techniques are available, including flap surgery, which enables tissue to be moved from one anatomical location to another. Perforating skin/subcutaneous flaps are segments of skin and subcutaneous cellular tissue vascularized by a feeder vascular pedicle. This surgical technique has virtually zero donor-site morbidity, as it is no longer necessary to harvest muscle to ensure reliable vascularization of the flap.

Flap vascularization is a variable mechanism, complex to describe and understand. For cutaneous and subcutaneous (fatty) flaps, which account for the majority of flaps used, perforator flaps (vascularized by a subcutaneous perforator artery) have become the benchmark. Unfortunately, their vascularization is currently poorly understood, and depends on experimental work carried out on fresh cadaveric anatomical specimens. These cadaveric studies fail to take into account several key factors influencing perforasomes (perforasome: skin territory vascularized by a pedicle), namely body temperature, blood pressure, heart rate, intraoperative patient position and biological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70
* Reconstructive surgery using pedicled perforating flap or free perforating flap.
* Flap with a surface area of at least 50 cm2 (in order to have a sufficiently large surface area for good perfusion visualization)
* Pedicled perforating flaps group: Patients with pelvic eschar
* Free perforating flaps group: Traumatic pathology of the lower and/or upper limb

Exclusion Criteria:

* No consent obtained
* No social security affiliation
* Persons under court protection
* Persons participating in another study with an exclusion period still in progress

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
study the superficial tissue perfusion of flaps (flow speed) | Between Day -1 and Day +1 of surgery
  with PeriCam device
study the superficial tissue perfusion of flaps (flow speed) | Between Day -1 and Day +1 of surgery
  with PeriFlux device
study the superficial tissue perfusion of flaps (Infusion quality) | Between Day -1 and Day +1 of surgery
  with PeriCam device
study the superficial tissue perfusion of flaps (Infusion quality) | Between Day -1 and Day +1 of surgery
  with PeriFlux device
study the superficial tissue perfusion of flaps (Oxygenation quality) | Between Day -1 and Day +1 of surgery
  with PeriFlux device
study the superficial tissue perfusion of flaps (Colorimetric infusion quality scale) | Between Day -1 and Day +1 of surgery
  with PeriCam device

SECONDARY OUTCOMES:
study the superficial tissue perfusion of flaps (flow speed) | Between Day -1 and Day +3 of surgery
  with PeriCam device
study the superficial tissue perfusion of flaps (flow speed) | Between Day -1 and Day +3 of surgery
  with PeriFlux device
study the superficial tissue perfusion of flaps (flow speed) | Between Day -1 and Day +30 of surgery
  with PeriCam device
study the superficial tissue perfusion of flaps (flow speed) | Between Day -1 and Day +30 of surgery
  with PeriFlux device
study the superficial tissue perfusion of flaps (Infusion quality) | Between Day -1 and Day +3 of surgery
  with PeriCam device
study the superficial tissue perfusion of flaps (Infusion quality) | Between Day -1 and Day +3 of surgery
  with PeriFlux device
study the superficial tissue perfusion of flaps (Infusion quality) | Between Day -1 and Day +30 of surgery
  with PeriCam device
study the superficial tissue perfusion of flaps (Infusion quality) | Between Day -1 and Day +30 of surgery
  with PeriFlux device
study the superficial tissue perfusion of flaps (Oxygenation quality) | Between Day -1 and Day +3 of surgery
  with PeriFlux device
study the superficial tissue perfusion of flaps (Oxygenation quality) | Between Day -1 and Day +30 of surgery
  with PeriFlux device
study the superficial tissue perfusion of flaps (Colorimetric infusion quality scale) | Between Day -1 and Day +3 of surgery
  with PeriCam device
study the superficial tissue perfusion of flaps (Colorimetric infusion quality scale) | Between Day -1 and Day +30 of surgery
  with PeriCam device
Study the superficial tissue perfusion of flaps in relation to ultrasound exploration (flap perforating vessel flow) | Between Day -1 and Day +1 of surgery
Study the superficial tissue perfusion of flaps in relation to clinical observations (skin recoloration time) | Between Day -1 and Day +1 of surgery
Number of participants with signs of tissue suffering (delayed capillary refill, color change, skin breakdown, blister) as observed on clinical examination | Between Day -1 and Day +1 of surgery
  Clinical signs of tissue suffering will be recorded based on predefined clinical criteria: capillary refill time > 3 seconds, local discoloration (pallor or cyanosis), or cutaneous ulceration or blisters. These signs will be assessed by a trained plastic surgeon and documented on standardized observation forms.
Study the superficial tissue perfusion of flaps in relation to clinical observations ( scarring). | Between Day -1 and Day +1 of surgery
  Scarification will be performed on the flap surface in the area suspected of tissue compromise, using a sterile needle to superficially scratch the skin. The assessment will document whether bleeding occurs at the site of scarification. If bleeding is present, it will be classified as: arterial bleeding (bright red), venous bleeding (dark red), no bleeding (indicative of dry necrosis or severe ischemia).

IPD SHARING:
Plan to Share IPD: Undecided